CLINICAL TRIAL: NCT05088421
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study of the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of BWC0977 in Healthy Adult Volunteers
Brief Title: A First in Human Study of the Safety and Tolerability of Single and Multiple Doses of BWC0977 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bugworks Research Inc. (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C001-2020-01
Record Dates: First submitted 2021-09-09; First posted 2021-10-21 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Infectious Diseases; Bacterial Infections
Keywords: Safety; Tolerability; Pharmacokinetics; BWC0977
MeSH Terms: conditions — Communicable Diseases; Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, combined single and multiple ascending dose (SAD and MAD) trial
Who Masked: Participant, Investigator
Masking Description: Participants will be randomized in a 3:1 ratio of BWC0977 and Placebo. The following controls will be employed to maintain the double-blind status of the study Infusion solution containing active drug and placebo will be indistinguishable in appearance Randomization list will be provided to the study center pharmacist for dispensing purposes and kept in the pharmacy, accessible to the pharmacist and authorized personnel only PK results for the interim analyses between cohorts will be presented in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BWC0977 (Experimental): SAD Cohorts: Subjects will receive single doses of BWC0977 via IV infusion over 2 hours. Planned doses to be studied are 120, 240, 480, 720, and 1050mg.
  MAD Cohorts: Subjects will receive multiple doses of 240mg TID 7 days, 350mg TID 7 days BWC0977 via IV infusion over 2 hours in the first 2 cohorts. The dose for the B3 cohort will be determined based on safety and tolerability data from the previous two cohorts Up to three dose groups will be studied.
  Interventions: Drug: BWC0977
- Placebo (Placebo Comparator): Compounded solution minus BWC0977 The placebo used during this study is 5% Dextrose for injection. SAD Cohorts: Subjects will receive single infusions of placebo (Compounded solution minus BWC0977) over two hour.
  MAD Cohorts: Subjects will receive multiple infusions of placebo over 2 hour for 10 consecutive days. Frequency of infusions will be determined based on safety, tolerability and PK data obtained for BWC0977 in SAD Cohorts.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BWC0977 — SAD Cohorts: Double-blind dosing will occur. Six participants will receive single doses of BWC0977. The dose escalation steps may be altered following review of the safety data upon completion of each cohort.
  MAD Cohorts: Double blind dosing will occur. Six participants in each cohort will receive multiple doses of BWC0977. The dose escalation steps may be altered following review of the safety data upon completion of each cohort. Dosing will commence on the morning of Day 1. Dosing frequency to be confirmed based on safety, tolerability and PK data from SAD cohorts. Daily dosing will continue for a total of 10 consecutive days.
  Arms: BWC0977
Drug: Placebo — SAD Cohorts: Two participants in each cohort will receive matching placebo. MAD Cohorts: Two participants in each cohort will receive matching placebo.
  Other Names: Compounded solution minus BWC0977
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of single and multiple intravenous doses of BWC0977 when administered to healthy adult volunteers.

DETAILED DESCRIPTION:
This Phase 1 study is designed to assess the safety, tolerabilty and pharmcokinetics of single and multiple intravenous doses of BWC0977 when administered to healthy adult volunteers. This is a randomized double-blind, placebo-controlled, ascending dose, multi-cohort trial. A total of 64 healthy volunteers are expected to be enrolled into 8 Cohorts. The study will be conducted in two phases: A single ascending dose (SAD) phase, followed by a multiple ascending dose (MAD) phase. In SAD, participants in Cohorts 1 - 5 will receive one dose of BWC0977 or placebo. In MAD, participants in Cohorts 6 - 8 will receive multiple doses of BWC0977 or placebo for 10 consecutive days at a dose deemed safe and tolerable as determined in the preceding SAD Cohorts. In both parts sequential cohorts will be exposed to increasing doses of BWC0977.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be eligible for study participation:

1. Healthy male or female 18 to 55 years of age, inclusive, at time of consent.
2. Body mass index (BMI) ≥ 19.0 and ≤ 30.0 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive).
3. Medically healthy without clinically significant abnormalities at the screening visit or Day -1, including:

   1. No findings in Physical examination or vital signs (including temperature, heart rate, respiratory rate, and blood pressure) that the Principal Investigator (PI) determines would interfere with interpretation of study results.
   2. Electrocardiograms (ECGs) without clinically significant abnormalities, including a QT duration corrected for heart rate by Fridericia's formula (QTcF) interval duration ≤450 msec (for males), and ≤470 msec (for females) obtained as an average from the triplicate screening ECGs after at least 5 minutes in a supine quiet-rest position.
   3. Clinically significant abnormalities in the screening clinical laboratory tests, as determined by the Investigator. Repeat testing could be performed at the Investigator's discretion.
4. Willing

Exclusion Criteria:

Volunteers who meet any of the following criteria will be excluded from the study:

1. Women who are pregnant and/or nursing.
2. History or presence of significant cardiovascular (including QT prolongation, clinically significant hypokalemia, or other proarrhythmic conditions), pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine (including glucose intolerance, diabetes mellitus), immunologic (including asthma or seasonal allergies [that require intermittent use of steroids or other medication]), musculoskeletal (including tendinopathy), dermatologic, or neurological disease (including seizure disorders, psychiatric disorders), including any acute illness or surgery within the past 3 months determined by the PI to be clinically relevant.
3. A serum creatinine value on Day -1 (check-in) that increased by more than 0.2 mg/dL (or 15.25 µmol/L) from the Screening value.
4. History of photosensitivity to quinolones.
5. History of known or suspected Clostridium difficile infection.
6. Any condition that necessitated hospitalisation within the 3 months prior to Day -1 or is likely to require so during the study.
7. Positive test for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV antibodies), or human immunodeficiency virus antibody (antibodies to HIV-1, HIV-2) or tuberculosis (TB) at screening.
8. Exposure to any prescription medications (small molecules, biologics including vaccines) or, systemically administered OTC drugs, dietary supplements or herbal remedies, within 30 days or 5 half-lives (if known), whichever is longer, prior to Day -1. Discussion between the PI and the Sponsor Medical Monitor is encouraged regarding prior use of any medications during the pre-dose period.

   Note: An exception is made for hormonal contraceptives and a limited amount of paracetamol (a maximum of 4 doses per day of 500-mg paracetamol, and no more than 3 g per week) for the treatment of headache or any other pain.
9. Documented hypersensitivity reaction or anaphylaxis to any medication.
10. Smoker (including tobacco, e-cigarettes or marijuana) or nicotine user within 1 month prior to participation in the study
11. Positive urine drug/alcohol testing at screening or check-in (Day -1), or history of substance abuse or alcohol abuse (defined as greater than 2 standard drinks on average each and every day, where one standard drink is defined as containing 10 g of alcohol and is equivalent to 1 can or stubby of mid-strength beer, 30 ml nip spirits, or 100 ml wine) within the previous 5 years (may be repeated once per timepoint, at the discretion of the PI, in the instance of a positive result).
12. Donation of blood or plasma within 30 days prior to randomization, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of study enrollment.
13. Previous participation in this study or previous participation in another study within 5 half-lives (if known) of the agent, whichever is longer, of Day 1. Note: prior participation at any time in non-invasive methodology trials in which no drugs were given is acceptable.
14. Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pummelos, other citrus fruits, grapefruit hybrids or fruit juices containing such products from 7 days prior to the first dose of study medication.
15. Employee or family member of an employee of the Sponsor, CRU, or clinical research organization at which the study will be conducted.
16. Unable to cooperate fully with the requirements of the study protocol, including the schedule of assessments, or likely to be non-compliant with any study requirements.
17. Any disease or condition (medical or surgical) that, by the determination of the PI, precludes the subject's participation in the study or would place the subject at risk as a result of participation in the study.

Note: Volunteers should refrain from consumption of any foods containing poppy seeds within 48 hours (2 days) prior to screening and prior to Day -1 to avoid false positive drug screen results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Efforts will be made to randomize approximately equal numbers of males and females to either active or placebo in Part 1 and Part 2 (including both genders).
Enrollment: 44 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs and serious adverse events (SAEs) overall and by intensity (Safety and tolerability). | SAD: Up to 7 days; MAD: Up to 15 days.
  This outcome combines the measure of the number of participants experiencing adverse events (AEs), the nature and severity of those AEs and their relationship to the study treatment.

SECONDARY OUTCOMES:
AUC[0-t] of BWC0977 following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  Area under the plasma concentration curve from time zero to last time of quantifiable concentration (AUC[0-t]) of BWC0977 following single dose administration
AUC[0-inf]) of BWC0977 following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  AUC from time zero to infinity (AUC[0-inf]) of BWC0977 following single dose administration
AUC[0-8], AUC[0-12], AUC[0-24]) of BWC0977 following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  AUC from time zero to 8, 12, and 24 hours (AUC[0-8], AUC[0-12], AUC[0-24]) of BWC0977 following single dose administration
Cmax of BWC0977 following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  Maximum observed plasma concentration (Cmax) of BWC0977 following single dose administration
Cmax of BWC0977 following repeat dose administration | Day 1 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, and 8 hours post infusion start Days 5, 6, 7, 8, and 9: pre-dose Day 10 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours post infusion start
  Maximum observed plasma concentration (Cmax) of BWC0977 following repeat dose administration
Terminal half-life (T1/2) | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  Terminal half-life (T1/2) of BWC0977 following single dose administration
Systemic clearance (CL) following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  Systemic clearance (CL) of BWC0977 following single dose administration
Systemic clearance (CL) following repeat dose administration | Day 1 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, and 8 hours post infusion start Days 5, 6, 7, 8, and 9: pre-dose Day 10 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours post infusion start
  Systemic clearance (CL) of BWC0977 following repeat dose administration
Volume of distribution at steady state (Vdss) following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  Volume of distribution at steady state (Vdss) of BWC0977 following single dose
Mean residence time (MRT) following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  Mean residence time (MRT) of BWC0977 following single dose administration
Pre-dose (trough) concentration (Cτ) at the end of the dosing interval | Day 1 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, and 8 hours post infusion start Days 5, 6, 7, 8, and 9: pre-dose Day 10 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours post infusion start
  Pre-dose (trough) concentration (Cτ) at the end of the dosing interval of BWC0977 following repeat dose administration
Observed accumulation ratio following repeat dose administration | Day 1 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, and 8 hours post infusion start Days 5, 6, 7, 8, and 9: pre-dose Day 10 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours post infusion start
  Observed accumulation ratio (Ro) of BWC0977 following repeat dose administration
Volume of distribution at steady state following repeat dose administration | Day 1 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, and 8 hours post infusion start Days 5, 6, 7, 8, and 9: pre-dose Day 10 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours post infusion start
  Volume of distribution at steady state (Vdss) of BWC0977 following repeat dose

OTHER OUTCOMES:
Amount excreted in urine (Ae) following repeat dose administration | Day 1 pre-dose, 0-8 hours post infusion start Day 10: 0-8 hours post infusion start
  Amount excreted in urine (Ae) of BWC0977 following repeat dose administration
Amount excreted in urine (Ae) following single dose administration | Day 1 pre-dose, 0-2, 2-4, 4-8, 8-12, and 12-24 hours post infusion start
  Amount excreted in urine (Ae) of BWC0977 following single dose administration
Fraction of the dose excreted in urine (fe) following single dose administration | Day 1 pre-dose, 0-2, 2-4, 4-8, 8-12, and 12-24 hours post infusion start
  Fraction of the dose excreted in urine (fe) of BWC0977 following single dose administration
Fraction of the dose excreted in urine (fe) following repeat dose administration | Day 1 pre-dose, 0-8 hours post infusion start Day 10: 0-8 hours post infusion start
  Fraction of the dose excreted in urine (fe) of BWC0977 following repeat dose administration
Renal Clearance (CLr) following single dose administration | Day 1 pre-dose, 0-2, 2-4, 4-8, 8-12, and 12-24 hours post infusion start
  Renal Clearance (CLr) of BWC0977 following single dose administration
Renal Clearance (CLr) following repeat dose administration | Day 1 pre-dose, 0-8 hours post infusion start Day 10: 0-8 hours post infusion start
  Renal Clearance (CLr) of BWC0977 following repeat dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Angela Molga, MD, Principal Investigator — CMAX Clinical Research
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hameed P S, Kotakonda H, Sharma S, Nandishaiah R, Katagihallimath N, Rao R, Sadler C, Slater I, Morton M, Chandrasekaran A, Griffen E, Pillai D, Reddy S, Bharatham N, Venkatesan S, Jonnalagadda V, Jayaraman R, Nanjundappa M, Sharma M, Raveendran S, Rajagopal S, Tumma H, Watters A, Becker H, Lindley J, Flamm R, Huband M, Sahm D, Hackel M, Mathur T, Kolamunnage-Dona R, Unsworth J, Mcentee L, Farrington N, Manickam D, Chandrashekara N, Jayachandiran S, Reddy H, Shanker S, Richard V, Thomas T, Nagaraj S, Datta S, Sambandamurthy V, Ramachandran V, Clay R, Tomayko J, Das S, V B. BWC0977, a broad-spectrum antibacterial clinical candidate to treat multidrug resistant infections. Nat Commun. 2024 Sep 18;15(1):8202. doi: 10.1038/s41467-024-52557-2. PMID 39294149